CLINICAL TRIAL: NCT04231331
Title: Multicenter, Randomized, Double-blind, Placebo-controlled, Phase 3 Study to Assess the Efficacy of Ertugliflozin on Reduction of Mitral Regurgitation in Patients With Functional Mitral Regurgitation Secondary to Left Ventricular Dysfunction
Brief Title: Ertugliflozin for Functional Mitral Regurgitation
Acronym: EFFORT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Asan Medical Center (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Duk-Hyun Kang, Professor, Asan Medical Center
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2019-1690
Record Dates: First submitted 2020-01-14; First posted 2020-01-18 (Actual); Results first posted 2025-01-06 (Actual); Last update posted 2025-01-06 (Actual); Status verified 2024-11

CONDITIONS: Mitral Valve Insufficiency; Left Ventricular Systolic Dysfunction
MeSH Terms: conditions — Mitral Valve Insufficiency; Ventricular Dysfunction, Left | interventions — ertugliflozin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): All patients will receive placebo in addition to their usual medications. Titration of HF medications should be completed and patients must take a stable, optimized dose of a β-blocker and an ACE inhibitor (or ARB) for at least 4 weeks prior to study entry.
  Interventions: Drug: Placebo
- Ertugliflozin (Active Comparator): All patients will receive ertugliflozin 5 mg qd in addition to their usual medications. Titration of HF medications should be completed and patients must take a stable, optimized dose of a β-blocker and an ACE inhibitor (or ARB) for at least 4 weeks prior to study entry.
  Interventions: Drug: Ertugliflozin

INTERVENTIONS:
Drug: Ertugliflozin — Ertugliflozin 5mg qd for 12 months
  Other Names: Steglatro
  Arms: Ertugliflozin
Drug: Placebo — Placebo qd for 12 months
  Arms: Placebo

SUMMARY:
In patients with heart failure (HF) and left ventricular (LV) dilation, adverse LV remodeling causes tethering of mitral valve (MV) preventing sufficient coaptation of normal leaflets and resulting in functional MR. Because secondary functional MR usually develops as a result of LV dysfunction, guideline-directed medical therapy for HF forms the mainstay of therapy. However, beta blockers, angiotensin-converting-enzyme (ACE) inhibitors, and angiotensin receptor blockers (ARB) fail to reverse adverse LV remodeling and functional MR, and the morbidity and mortality of patients with functional MR remain high despite standard medical therapy. Randomized trials to explore cardiovascular (CV) benefit of the sodium-glucose co-transporter-2 (SGLT2) inhibitor have been performed and showed a significant reduction on the risk of CV death or hospitalization for HF. However, its effect on cardiac structure and function was not evaluated and further mechanistic studies are needed to interpret beneficial clinical effects of the SGLT2 inhibitors. Based on studies demonstrating SGLT2 inhibitors' favorable effects on LV modeling, investigators hypothesize that SGLT2 inhibitor, ertugliflozin, is effective on improving MR in patients with functional MR secondary to LV dysfunction and try to examine this hypothesis in a multicenter, double-blind, randomized comparison study using echocardiography.

DETAILED DESCRIPTION:
In patients with heart failure (HF) and left ventricular (LV) dilation, adverse LV remodeling causes tethering of mitral valve (MV) preventing sufficient coaptation of normal leaflets and resulting in functional MR. Because secondary functional MR usually develops as a result of LV dysfunction, guideline-directed medical therapy (GDMT) for HF forms the mainstay of therapy. However, beta blockers, angiotensin-converting-enzyme (ACE) inhibitors, and angiotensin receptor blockers (ARB) fail to reverse adverse LV remodeling and functional MR, and the morbidity and mortality of patients with functional MR remain high despite standard medical therapy. A recent randomized trial (COAPT) proved that reduction of functional MR by transcatheter MV repair resulted in a lower rate of hospitalization for HF and lower mortality in patients with HF and significant secondary MR, but more than two-thirds of such patients either died or were hospitalized for HF within 5 years. Thus, optimization of GDMT for timely reduction of functional MR is important, because the persistence of severe functional MR despite GDMT contributes to a vicious cycle of deterioration and leads to irreversible LV dysfunction and a poorer prognosis.

Sodium-glucose co-transporter-2 (SGLT2) inhibitors reduce cardiac preload and afterload by natriuresis and lowering arterial stiffness, similar to the neprilysin inhibitor that facilitates sodium excretion and has vasodilating effects. Randomized trials to explore cardiovascular (CV) benefit of the SGLT2 inhibitor have been performed and showed a significant reduction on the risk of CV death or hospitalization for HF. Based on remarkable outcomes of recent clinical trials, SGLT2 inhibitors are recommended for HF with reduced EF and can be beneficial in HF with preserved EF. These outcome trials of SGLT2 inhibitors did not examine their effects on cardiac structure and function, and small imaging trials reported conflicting results in terms of the effect of a SGLT2 inhibitor on LV remodeling in patients with HFrEF and diabetes. Despite current recommendations of SGLT2 inhibitors for HF, SGLT2 inhibitors are rarely used in patients with HF with functional MR, as shown in the COAPT trial, because their effects on cardiac remodeling and functional MR are uncertain. The EFFORT trial (Ertugliflozin for Functional Mitral Regurgitation) was designed to evaluate the therapeutic efficacy of the SGLT2 inhibitor, ertugliflozin, on functional MR. The major hypothesis of this trial was that ertugliflozin would be superior to placebo in reducing functional MR associated with HF with mildly or moderately reduced EF.

ELIGIBILITY:
Inclusion Criteria:

* Patients must agree to the study protocol and provide written informed consent
* Outpatients ≥ 20 years of age, male or female
* Non-diabetic or type2 DM patients with HbA1c 7.0-10.5%
* Patients with secondary functional MR (stage B and C) and LV dysfunction

  * Symptoms due to coronary ischemia or heart failure may be present but symptoms due to MR should be absent
  * Normal mitral valve leaflets and chords
  * Regional or global wall motion abnormalities with mild or severe tethering of leaflet
  * MR whose ERO > 0.10 cm2 and which lasted > 6 months under medical treatment with a β-blocker and an ACE inhibitor (or ARB)
  * 35% < LV ejection fraction < 50%
* Dyspnea of NYHA functional class II or III
* Titration of HF medications should be completed and patients must take a stable, optimized dose of a β-blocker and an ACE inhibitor (or ARB) for at least 4 weeks prior to study entry

Exclusion Criteria:

* History of hypersensitivity or allergy to the study drug, drugs of similar chemical classes, or SGLT-2 as well as known or suspected contraindications to the study drug
* Current use or prior use of a SGLT-2 inhibitor or combined SGLT-1 and 2 inhibitor
* Known history of angioedema
* Any evidence of structural mitral valve disease, including prolapse of mitral leaflets and rupture of chords or papillary muscles
* Current acute decompensated heart failure or dyspnea of NYHA functional class IV
* Medical history of hospitalization within 6 weeks
* Symptomatic hypotension and/or a SBP < 100 mmHg at screening
* Estimated GFR < 45 mL/min/1.73m2
* History of ketoacidosis
* Evidence of hepatic disease as determined by any one of the following: AST or ALT values exceeding 2 x upper limit of normal (ULN) at screening visit (Visit 0), history of hepatic encephalopathy, history of esophageal varices, or history of portacaval shunt.
* Acute coronary syndrome, stroke, major CV surgery, PCI within 3 months
* Substantial myocardial ischemia requiring coronary revascularization, a plan of coronary revascularization or mitral valve intervention within 1 year
* Indication of cardiac resynchronization therapy, a plan of heart transplantation or implantation of cardiac resynchronization therapy
* History of severe pulmonary disease
* Significant aortic valve disease
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using a barrier method plus a hormonal method
* Pregnant or nursing (lactating) women
* Any clinically significant abnormality identified at the screening visit, physical examination, laboratory tests, or electrocardiogram which, in the judgment of the investigator, would preclude safe completion of the study

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2020-11-04 (Actual); Primary Completion 2023-11-15 (Actual); Study Completion 2023-11-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: DUK HYUN KANG, MD, Principal Investigator — Asan Medical Center
Locations (3):
- South Korea (3):
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Kang DH, Park SJ, Shin SH, Hwang IC, Yoon YE, Kim HK, Kim M, Kim MS, Yun SC, Song JM, Kang SM. Ertugliflozin for Functional Mitral Regurgitation Associated With Heart Failure: EFFORT Trial. Circulation. 2024 Jun 11;149(24):1865-1874. doi: 10.1161/CIRCULATIONAHA.124.069144. Epub 2024 May 1. PMID 38690659

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Analyses followed the intention-to-treat principle, where all randomized patients were included in the group to which they were originally allocated.
Period: Overall Study
Arm/Group | Placebo | Ertugliflozin
Started | 65 | 63
Completed | 56 | 58
Not Completed | 9 | 5

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Placebo
- Ertugliflozin: Ertugliflozin
- Total: Total of all reporting groups
Arm/Group | Placebo | Ertugliflozin | Total
Number analyzed (Participants) | 65 | 63 | 128
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 50 | 50 | 100
  >=65 years | 15 | 13 | 28
Age, Continuous [Mean (Standard Deviation); unit: years] | 67 (11) | 65 (12) | 66 (11)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 27 | 23 | 50
  Male | 38 | 40 | 78
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Diabetes [Count of Participants; unit: Participants] | 9 | 7 | 16
Atrial fibrillation [Count of Participants; unit: Participants] | 32 | 33 | 65

OUTCOME MEASURES:

1. Primary Outcome: Change of EROA
Description: Change of effective regurgitant orifice area (EROA) of functional mitral regurgitation
Time Frame: Baseline and 12 months
Population: Primary analysis included all 114 patients who completed the study.
Measure: Mean (Standard Deviation); unit: square cm
Arm/Group | Placebo | Ertugliflozin
Number analyzed (Participants) | 56 | 58
square cm | 0.03 (0.12) | -0.05 (0.06)
Statistical Analysis 1: Comparison: Placebo vs Ertugliflozin; Based on our previous study, we assumed a common baseline mean EROA of 0.21 cm2 with a common standard deviation of 0.11 cm2. Given these assumptions, we calculated that a sample size of 204 patients randomly assigned to two groups, would provide 90% power to detect a difference of 0.05 cm2 in the EROA between the ertugliflozin and placebo groups, using a two-sided t test with an alpha level of 0.05; Test type: Superiority; p < 0.001, t-test, 2 sided — P-value <0.05 was considered statistically significant

2. Secondary Outcome: Change of Regurgitant Volume
Description: Change of regurgitant volume of functional mitral regurgitation
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: mL
Arm/Group | Placebo | Ertugliflozin
Number analyzed (Participants) | 56 | 58
mL | 39.3 (31.1) | 24.6 (14.3)

3. Secondary Outcome: Change of End-systolic Volume Index
Description: Left ventricular end-systolic volume was measured with the use of echocardiography. Left ventricular end-systolic volume index was obtained by dividing end-systolic volume by body surface area.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: mL/square m
Arm/Group | Placebo | Ertugliflozin
Number analyzed (Participants) | 56 | 58
mL/square m | -3.6 (13.4) | -4.1 (8.1)

4. Secondary Outcome: Change of End-diastolic Volume Index
Description: Left ventricular end-diastolic volume was measured with the use of echocardiography. Left ventricular end-diastolic volume index was obtained by dividing end-diastolic volume by body surface area.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: mL/square m
Arm/Group | Placebo | Ertugliflozin
Number analyzed (Participants) | 56 | 58
mL/square m | -5.7 (17.2) | -4.7 (11.0)

5. Secondary Outcome: Change of NT-proBNP
Description: Change of NT-proBNP (N-terminal of the prohormone brain natriuretic peptide)
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: pg/mL
Arm/Group | Placebo | Ertugliflozin
Number analyzed (Participants) | 56 | 58
pg/mL | 126 (1112) | -154 (815)

6. Secondary Outcome: Change of Left Ventricular Global Longitudinal Strain
Description: Myocardial strain is a measure of percenage shortening of myocardium. Myocardial strain measurement was performed with a semiautomated alogithm using speckle-tracking echocardiogrphy. Measurements of eft ventricular global longitudinal strain were made in the 3 standard apical views and averaged.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: percent change of myocardial length
Arm/Group | Placebo | Ertugliflozin
Number analyzed (Participants) | 56 | 58
percent change of myocardial length | 0.10 (2.68) | -1.34 (2.57)

7. Secondary Outcome: Change of LA End-systolic Volume Index
Description: Left atrial end-systolic volume was measured with the use of echocardiography. Left atrial end-systolic volume index was obtained by dividing end-systolic volume by body surface area.
Time Frame: Baseline and 12 months
Measure: Mean (Standard Deviation); unit: mL/square m
Arm/Group | Placebo | Ertugliflozin
Number analyzed (Participants) | 56 | 58
mL/square m | 3.2 (17.7) | -2.8 (13.8)

ADVERSE EVENTS:
Time Frame: 12 months
Arm/Group | Placebo | Ertugliflozin
All-Cause Mortality (participants affected / at risk) | 3/65 | 0/63
Serious Adverse Events (participants affected / at risk) | 3/65 | 1/63
Other Adverse Events (participants affected / at risk) | 0/65 | 0/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=65) | Ertugliflozin (N=63)
Heart failure hospitalization (Cardiac disorders) | 3 (3) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Placebo (N=65) | Ertugliflozin (N=63)
Heart failure hospitalization (Cardiac disorders) | 0 (0) | 0 (0)

LIMITATIONS AND CAVEATS:
Because enrollment of trial patients was affected by the COVID-19 pandemic, the present trial did not reach the calculated sample size.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-05-22): https://cdn.clinicaltrials.gov/large-docs/31/NCT04231331/Prot_SAP_000.pdf